CLINICAL TRIAL: NCT03842241
Title: Changes of Kinematics, Muscle Activity, Joint Contact Force of Foot Orthoses for Individual of Flat Foot After Functional Fatigue Protocol
Brief Title: Effects of Fatigue and Foot Orthoses on Lower Extremity EMG and Biomechanics for Individuals With Flat Foot
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: YM107091E
Record Dates: First submitted 2019-01-17; First posted 2019-02-15 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2019-02

CONDITIONS: Flexible Flatfoot
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- WIth foot orthoses: Device: Non-custom made foot orthoses
  Interventions: Device: Non-custom made foot orthoses
- Without foot orthoses: Other: without foot orthoses

INTERVENTIONS:
Device: Non-custom made foot orthoses — Foot orthoses is an orthotic devices which are used to support arch and rear-foot and put it in a good alignment.
  Groups: WIth foot orthoses

SUMMARY:
Determine the effects of non-custom made foot orthoses on the kinematics, muscle activity and joint contact force after fatigue and compare the rate of fatigue in flexible flat foot with and without foot orthoses

ELIGIBILITY:
Inclusion Criteria:

* Bilateral flexible flatfoot( navicular bone drop greater than 10 mm)

Exclusion Criteria:

* History of foot and ankle surgery, inflammatory joint disease
* History of lower extremity injury in six months
* Known pathological or neurological disorders that could affect gait pattern

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Flexible flatfoot
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Lower extremities kinetic | 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed, after one week, 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed
  Three dimensional motion data were collected using a Vicon camera system during walking.
  Using motion capture system data to calculate the hip, knee internal/external rotation moment and ankle inversion/eversion moment via inverse dynamics method.
Peak and average amplitude during stance phase | 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed, after one week, 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed
  EMG data were collected using a Delsys, and Biopac EMG system during walking. Tibialis anterior/Peroneal longus/Abductor hallucis longus muscle activity were measured by electromyography (EMG).
Lower extremities kinematic | 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed, after one week, 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed
  Lower limbs alignment, including hip, knee and ankle joints. Using motion capture system data to calculate the joint angles.

SECONDARY OUTCOMES:
Lower extremities kinematic | 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed, after one week, 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed
  Three dimensional kinematics were collected using a Vicon camera system during walking.
  Lower limbs alignment, including hip, knee and ankle joints. Using motion capture system data to calculate the joint angles.
Peak and average amplitude during stance phase | 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed, after one week, 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed
  EMG data were collected using a Delsys, and Biopac EMG system during walking. Medial gastrocnemius/Rectus femoris/Bicep femoris muscle activity were measured by EMG.
Time of completed fatigue protocols | 1 minutes after fatigue protocol completed
  Time of completed the course will be recorded.
Inter-joint contact force | 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed, after one week, 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed
  Hip, knee ,and ankle inter-joint contact force: Anybody modeling system is used to model the inter-joint contact force
Lower extremities kinetic | 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed, after one week, 10 minutes before fatigue protocol start, 5 minutes after fatigue protocol completed
  Three dimensional motion data were collected using a Vicon camera system during walking.
  Using motion capture system data to calculate the hip, knee flexion/extension, adduction/abduction moment and ankle dorsiflexion/plantarflexion, and adduction/abduction moment via inverse dynamics method.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan